CLINICAL TRIAL: NCT03525457
Title: Response to Non Surgical Periodontal Therapy in a Chronic Kidney Disease Population Candidates to Kidney Transplant
Brief Title: Response to Periodontal Therapy in a Chronic Kidney Disease Population
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Pontificia Universidad Catolica de Chile (Other)
Responsible Party: Principal Investigator, Maité Souyet, DDS, MsC, Pontificia Universidad Catolica de Chile
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 180104004
Record Dates: First submitted 2018-05-02; First posted 2018-05-15 (Actual); Last update posted 2018-08-31 (Actual); Status verified 2018-08

CONDITIONS: Chronic Kidney Disease Stage 5; Periodontal Disease
Keywords: Glomerular filtration rate; Periodontitis; Chronic kidney disease
MeSH Terms: conditions — Renal Insufficiency, Chronic; Periodontal Diseases; Periodontitis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Non surgical periodontal therapy
  Interventions: Procedure: Non Surgical Periodontal Therapy

INTERVENTIONS:
Procedure: Non Surgical Periodontal Therapy — Non Surgical Periodontal Therapy in 2 to 3 sessions

SUMMARY:
This study will evaluate periodontal and systemic parameters of a cohort of chronic kidney disease (stage 5) patients, before and three months after non-surgical periodontal treatment. It does not consider a control group.

DETAILED DESCRIPTION:
Dental biofilm is a source of inflammation and infection of periodontal tissues. In the last 20 years the interaction between periodontal infections and systemic conditions has been largely studied, suggesting that the inflammation caused in the periodontal tissues could cause a response in other parts of the body.

Recent studies suggest that there could be an association between periodontal disease and chronic kidney disease.

ELIGIBILITY:
Inclusion Criteria:

* Chronic kidney disease patients in Stage 5 (candidates to renal transplant)

Exclusion Criteria:

* Younger than 18 year old.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 65 (Estimated)
Dates: Start 2018-08-06 (Actual); Primary Completion 2019-08 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Change in Clinical Attachment Level (CAL) | 3 months
  Change from baseline CAL (in mm) at three months

SECONDARY OUTCOMES:
Change in Bleeding on probing (BOP) | 3 months
  Change from baseline BOP (%) at three months

CONTACTS AND LOCATIONS:
Overall Officials: Maite C Souyet, MsC, Principal Investigator — Pontificia Universidad Catolica de Chile
Locations (1):
- Clínica Odontológica Docente UC, Santiago, Santiago Metropolitan, Chile

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Almeida S, Figueredo CM, Lemos C, Bregman R, Fischer RG. Periodontal treatment in patients with chronic kidney disease: a pilot study. J Periodontal Res. 2017 Apr;52(2):262-267. doi: 10.1111/jre.12390. Epub 2016 May 2. PMID 27135778
- [Background] Graziani F, Cei S, La Ferla F, Vano M, Gabriele M, Tonetti M. Effects of non-surgical periodontal therapy on the glomerular filtration rate of the kidney: an exploratory trial. J Clin Periodontol. 2010 Jul;37(7):638-43. doi: 10.1111/j.1600-051X.2010.01578.x. Epub 2010 May 25. PMID 20500539
- [Background] Chambrone L, Foz AM, Guglielmetti MR, Pannuti CM, Artese HP, Feres M, Romito GA. Periodontitis and chronic kidney disease: a systematic review of the association of diseases and the effect of periodontal treatment on estimated glomerular filtration rate. J Clin Periodontol. 2013 May;40(5):443-56. doi: 10.1111/jcpe.12067. Epub 2013 Feb 21. PMID 23432795
- [Background] Limeres J, Garcez JF, Marinho JS, Loureiro A, Diniz M, Diz P. Early tooth loss in end-stage renal disease patients on haemodialysis. Oral Dis. 2016 Sep;22(6):530-5. doi: 10.1111/odi.12486. Epub 2016 May 27. PMID 27038430